CLINICAL TRIAL: NCT04900415
Title: Olfactory and Neurosensory Rehabilitation in Coronavirus 2019 (COVID-19)-Related Olfactory Dysfunction (OD)
Brief Title: Olfactory and Neurosensory Rehabilitation in COVID-19-related Olfactory Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ivan FN Hung MD (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Sponsor-Investigator, Ivan FN Hung MD, Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 20-454
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Coronavirus Disease 2019
Keywords: Vitamin A; Smell training; COVID-19; Olfactory dysfunction; Anosmia; Functional MRI
MeSH Terms: conditions — COVID-19; Anosmia | interventions — Vitamin A

STUDY DESIGN:
Intervention Model Description: Patients with prolonged COVID-19-related olfactory dysfunction will be assigned to the intervention (group A or B) or control (group C) arms:
  Intervention arm A. 14-day course of daily oral vitamin A 7500µg RAE (retinol activity equivalents) in combination with smell training three times per day for 4 weeks; or B. Smell training three times per day for 4 weeks alone; or
  Control arm C. Observation
Who Masked: Investigator, Outcomes Assessor
Masking Description: All study participants will receive baseline and follow up resting-state functional (rs-fMRI) brain scans during the study period. The radiologists assessing and analysing the rs-fMRI images will be blinded to the treatment regimens received by the study subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin A and smell training (Experimental): 14-day course of daily oral vitamin A 7500µg RAE in combination with smell training three times per day for 4 weeks
  Interventions: Drug: Vitamin A; Device: Electronic portable aromatic rehabilitation (EPAR) diffuser
- Smell training (Active Comparator): Smell training three times per day for 4 weeks
  Interventions: Device: Electronic portable aromatic rehabilitation (EPAR) diffuser
- Control (No Intervention): Observation

INTERVENTIONS:
Drug: Vitamin A — Metabolic supplement for neurogenesis at the olfactory apparatus
  Arms: Vitamin A and smell training
Device: Electronic portable aromatic rehabilitation (EPAR) diffuser — Handheld essential oil ultrasonication diffuser technology
  Arms: Smell training; Vitamin A and smell training

SUMMARY:
A combination of oral vitamin A (VitA) and intense aromatic chemosensory smell training (ST) by pulse aromatic stimulation will expedite the neurosensory recovery of olfaction in patients suffering from prolonged COVID-19-related olfactory dysfunction (OD).

DETAILED DESCRIPTION:
This is an open-labeled randomised-controlled trial (RCT) investigating the safety and therapeutic efficacy of oral VitA in combination with ST for patients suffering from prolonged COVID-19-related OD.

Prior to the initiation of treatment, all patients will receive subjective and objective olfactory assessments. Comprehensive ear, nose, and throat (ENT) examination will be performed to rule out alternative causes of OD. All participants will receive resting-state functional magnetic resonance imaging (rs-fMRI) of the brain before treatment as baseline evaluation.

Patients with prolonged COVID-19-related OD will be assigned to the intervention (group A or B) or control (group C) arms:

Intervention arm A. 14-day course of daily oral VitA 7500µg RAE (retinol activity equivalents) in combination with ST three times per day for 4 weeks; or B. ST three times per day for 4 weeks alone; or

Control arm C. Observation

In addition, healthy controls who were tested negative for SARS-CoV-2 by reverse transcription polymerase chain reaction (RT-PCR) will receive rs-fMRI brain scans for radiological comparisons.

At the completion of the trial, subjective and objective olfactory assessments will be repeated to document clinical changes in olfaction. Follow-up rs-fMRI will be performed to document neuroradiological changes in the brain structures and cerebral network functional connectivity (FC).

ELIGIBILITY:
Inclusion Criteria:

1. Adult out-patient (≥18 years of age)
2. Previously diagnosed with coronavirus disease 2019 (COVID-19) by laboratory confirmation using reverse transcriptase polymerase chain reaction (RT-PCR) for the detection of severe acute respiratory virus coronavirus 2 (SARS-CoV-2)
3. Complaints of persistent olfactory disturbances, subjectively
4. Quantitatively documented to have olfactory dysfunction by

   1. Butanol threshold test (BTT)
   2. Smell identification test (SIT)
5. All subjects give written informed consent
6. Subjects must be available to complete the study and comply with study procedures.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures
2. Allergy or severe reactions to the study drug or smell training
3. Pregnant or breastfeeding women
4. Pre-existing factors which may account for persistent olfactory dysfunction besides COVID-19 (e.g. nasal polyps, obstructive lesions within the nasal cavity, severe anatomical malformations…)
5. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.
6. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Subjective olfactory assessment | 4 weeks
  Subjective olfactory assessment by the Sino-Nasal Outcome Test (SNOT-22).
Objective olfactory assessment by the butanol threshold test (BTT) | 4 weeks
  Objective measurements of olfactory sensitivity, as determined by the detection of different concentrations of butanol.
Objective olfactory assessment by the smell identification test (SIT) | 4 weeks
  Objective categorization of olfactory status by the smell identification test (SIT).

SECONDARY OUTCOMES:
Interim neuroradiological changes after 2 weeks of olfactory treatment | 2 weeks
  Group independent component (GIC) and cerebral network functional connectivity (FC) analyses of the olfactory, gustatory, somatosensory, and integrative networks using rs-fMRI scans, before and at 2 weeks after olfactory treatment in COVID-19 patients with olfactory dysfunction (OD)
Neuroradiological changes after olfactory treatment at the end of study | 4 weeks
  Group independent component analyses and functional connectivity analyses of the olfactory, gustatory, somatosensory, and integrative networks by resting-state functional MRI brain scans, before and after treatment in COVID-19 patients with olfactory dysfunction at 4 weeks.
Interim neuroradiological changes after oral vitamin A in combination with smell training versus smell training alone | 2 weeks
  Group independent component analyses and functional connectivity analyses of the olfactory, gustatory, somatosensory, and integrative networks by resting-state functional MRI brain scans, between combined VitA and smell training (ST) versus ST alone in COVID-19 patients with olfactory dysfunction at 2 weeks.
Neuroradiological brain changes in the intervention group versus observation group at the end of study | 4 weeks
  Group independent component analyses and functional connectivity analyses of the olfactory, gustatory, somatosensory, and integrative networks by resting-state functional MRI brain scans, in the interventional versus control arms (observation) in COVID-19 patients with olfactory dysfunction at 4 weeks.
Neuroradiological brain changes in the intervention group versus healthy control group at the end of study | 4 weeks
  Group independent component analyses and functional connectivity analyses of the olfactory, gustatory, somatosensory, and integrative networks by resting-state functional MRI brain scans, in COVID-19 patients with olfactory dysfunction compared with healthy controls at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - The University of Hong Kong, Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No